CLINICAL TRIAL: NCT04093401
Title: An Open-Label, Single Blind Study of How Knowledge of Risk of Subsequent Basal Cell Carcinoma Affects Compliance With Requested Follow-Up in Patients With First Basal Cell Carcinoma
Brief Title: The VIDYA Study-designed to Determine if Patients With a History of Basal Cell Carcinoma Are More Inclined to Return for Follow-up if Their Risk of a Subsequent Basal Cell Carcinoma is Quantitated.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW19002; 2019-0077 (Other: Institutional Review Board); A534300 (Other: UW Madison); SMPH/DERMATOLOGY/DERMATOLOG (Other: UW Madison)
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects will be assigned to the control arm if their subject ID is an odd number. Control arm subjects will not receive counseling for individualized risk assessment for developing a second basal cell carcinoma.
- Individualized risk assessment (Experimental): Subjects will be assigned to the intervention arm (i.e., informed of their individualized risk assessment) if their subject ID is an even number. Subjects in the intervention arm will be informed of their estimated 1-year, 3-year, and 5-year risk of developing a second basal cell carcinoma.
  Interventions: Other: individualized risk assessment

INTERVENTIONS:
Other: individualized risk assessment — Individualized risk assessment of developing a second basal cell carcinoma
  Arms: Individualized risk assessment

SUMMARY:
While current guidelines call for annual follow-up for patients with a history of basal cell carcinoma, compliance with these guidelines is imperfect. It is hypothesized that if patients are informed of the quantitative risk of a subsequent basal cell carcinoma based on individualized risk factors, the compliance rate for follow-up will improve.

The primary objective of this study is to assess one-year compliance with requested follow-up for patients with recent history of basal cell carcinoma, among those who receive standard sun avoidance counseling and request for follow-up compared to those who receive, in addition, an estimate of their mathematical risk of a subsequent basal cell carcinoma based on individualized risk factors.

DETAILED DESCRIPTION:
This is an open-label, single-blind study to evaluate the effect of informing subjects of their individualized risk of a subsequent basal cell carcinoma on proportion of subjects who achieve compliance with requested follow-up with a dermatology healthcare provider, defined as in-person follow-up within 365 days following diagnosis of initial basal cell carcinoma.

Subjects will be randomized 1:1 to "intervention" (knowledge of individualized risk) or "control" (lack of awareness of individualized risk). Investigators will be aware of the modelled risk of a subsequent basal cell carcinoma for all subjects, but only subjects randomized to the "intervention" arm will be informed of their modelled risk. All subjects will receive standard sun avoidance counseling and will be requested to follow-up no later than 365 days from initial basal cell carcinoma diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed with at least one Basal Cell Carcinoma within 30 days prior to enrollment
* Able and willing to answer all questions accurately in the Individualized Risk Assessment

Exclusion Criteria:

* History of Basal Cell Carcinoma 31 or more days prior to enrollment
* Solid Organ Transplant Recipient
* History of Immunodeficiency (e.g., HIV infection, AIDS, genetic immunodeficiency
* Prisoner
* Psychiatric inpatients or people who are institutionalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have a followup second skin exam by a dermatologist within 1 year of diagnosis of their first basal cell carcinoma (BCC) | up to 13 months
  Number of participants who have a followup second skin exam by a dermatologist within 1 year of diagnosis of their first basal cell carcinoma (BCC)

SECONDARY OUTCOMES:
Frequency of sunscreen use when out in sun | up to 13 months
  Frequency of sunscreen use when out in sun Participants will be instructed to use sunscreen on a daily basis during April - October. Regularity of sunscreen use will be queried during sunny parts of the year (spring to fall). Frequency of sunscreen use will be measured as daily use during the months of April - October
Frequency of sunburns within the past year | up to 13 months
  Frequency of sunburns within the past year

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Glinert, MD, Principal Investigator — clinical professor

IPD SHARING:
Plan to Share IPD: No